CLINICAL TRIAL: NCT00592722
Title: A Multi-Centre Clinical Study in Chronic Spinal Cord Injury Patients
Status: Completed | Type: Observational
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Director, Clinical Trial Centre, The University of Hong Kong
Other Study IDs: CN100b
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish a solid foundation, e.g. network and a coordinating centre for testing new SCI therapies in forthcoming randomized controlled multi-centre clinical trials following international standards and guidelines

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects, 18 to 60 years of age;
2. Have a clinical diagnosis of chronic SCI (defined as a history of ≥ 12 months suffering SCI);
3. The diagnosis of SCI was confirmed by MRI; and
4. Voluntarily signs and dates an Informed Consent Form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to any study-specific procedures

Exclusion Criteria:

1. Severe head injury;
2. Is medically or mentally unstable according to the judgement of the Investigator;
3. History of Multiple Sclerosis or peripheral demyelinating disease;
4. Likely to have experimental therapy;
5. Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The primary study outcomes will be the subject recruitment rate, the subject drip out rate, the number of missing values and the number of submitted incorrect values | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wise Young, MD, PhD, Study Director — The University of Hong Kong
Locations (5):
- China (3):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - 301 Orthopedic Hospital, Beijing
  - Second Affiliated Hospital of Third Military Medcial University, Chongqing
- Taiwan (2):
  - Buddhist Tzu Chi General Hospital, Hualien City
  - China Medical University Hospital, Taichung